CLINICAL TRIAL: NCT03248648
Title: Efficacy of Intra-articular Neostigmine Versus Ketamine for Postoperative Analgesia in Arthroscopic Knee Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Ghada Mohammed AboelFadl (Unknown); Abualauon Elbiblawy (Unknown)
Responsible Party: Principal Investigator, Amani Hassan Abdel-Wahab, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00008788
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Neostigmine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine group (Active Comparator): At the end of the surgery patients receive 0.5mg/dose neostigmine +18ml 0.25%bupivacaine in a total volume of 20 ml.
  Interventions: Drug: Neostigmine
- ketamine group (Active Comparator): At the end of the surgery patients receive 0.5 mg/kg ketamine+18ml 0.25%bupivacaine in a total volume of 20 ml.
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: Neostigmine — patient receive 0.5mg/dose neostigmine +18ml 0.25%bupivacaine in a total volume of 20 ml.
  Other Names: epistigmine
  Arms: Neostigmine group
Drug: ketamine — patient receive 0.5 mg/kg ketamine+18ml 0.25%bupivacaine in a total volume of 20 ml.
  Other Names: Ketalar
  Arms: ketamine group

SUMMARY:
To compare the efficacy of intra-articular administration of neostigmine versus ketamine as adjuvant analgesics after knee arthroscopy.

DETAILED DESCRIPTION:
Arthroscopic knee surgery is commonly performed as an outpatient procedure and is often associated with postoperative pain. Intraarticular (IA) local anesthetics (LA) are often used for prevention of pain after arthroscopic knee surgery; however, the degree of postoperative pain varies. In an effort to find the ideal regime for sufficient, long-lasting postoperative analgesia, many different drugs, including opioids, nonsteroidal anti-inflammatory drugs, ketamine, clonidine, and neostigmine, have been added to the IA LAs The investigators designed this study to compare the efficacy of intra-articular administration of neostigmine versus ketamine as adjuvant analgesics after knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* One hundred patients aged above 18-50 years (ASA I or II) scheduled for elective arthroscopic knee surgery under intrathecal anaesthesia will be enrolled in our study.

Exclusion Criteria:

* Absolute or relative contraindications for intrathecal anaesthesia,
* Allergy for the studied drugs.
* Patients having history of cardiovascular, cerebrovascular, and respiratory diseases,
* Patients receiving chronic pain treatment or hypertension treated with α methyldopa, clonidine or β adrenergic blockers were excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative analgesic consumption | 36 hours postoperative the total consumption of analgesics in the first 36h postoperative
  assessment of each patient on his bed at inpatient ward every 4 hours over a 36-hour period

SECONDARY OUTCOMES:
Postoperative visual analogue pain scale (VAS) | 36 hours postoperative
  assessment of each patient on his bed at inpatient ward every 4 hours over a 36-hour period

CONTACTS AND LOCATIONS:
Overall Officials: Abualauon Elbiplaoy, lectural of anesthesia, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided